CLINICAL TRIAL: NCT02065622
Title: A Double-Blind, Randomized, Multicenter Study of Higher Versus Standard Adalimumab Dosing Regimens for Induction and Maintenance Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Study to Evaluate the Safety and Efficacy of Two Adalimumab Dosing Regimens in Subjects With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-033; 2013-001682-16 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-09

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Induction (Main Study + Japan Sub-study): I-SD (Experimental): Induction Standard Dose: Double-blind adalimumab regimen of 160 mg at Week 0 followed by 80 mg at Week 2, 40 mg at Week 4, and 40 mg at Week 6.
  Interventions: Drug: Adalimumab; Other: Placebo
- Induction (Main Study + Japan Sub-study): I-HD (Experimental): Induction Higher Dose: Double-blind adalimumab regimen of 160 mg at Weeks 0, 1, 2, and 3 followed by 40 mg at Week 4, and 40 mg at Week 6.
  Interventions: Drug: Adalimumab
- Maintenance (Main Study + Japan Sub-study): M-SD (Experimental): Maintenance Standard Dose: Double-blind adalimumab 40 mg every other week (eow), for 44 weeks.
  Interventions: Drug: Adalimumab; Other: Placebo
- Maintenance (Main Study + Japan Sub-study): M-HD (Experimental): Maintenance Higher Dose: Double-blind adalimumab 40 mg every week (ew) for 44 weeks.
  Interventions: Drug: Adalimumab
- Maintenance (Main Study): TDM Regimen (Experimental): Double-blind adalimumab 40 mg eow at Week 8 and Week 10, with possible dose adjustments at Weeks 12, 24, and 37 based on criteria assessing blinded adalimumab serum concentration and rectal bleeding subscore (RBS) assessments.
  Interventions: Drug: Adalimumab; Other: Placebo

INTERVENTIONS:
Drug: Adalimumab
  Other Names: Humira
Other: Placebo
  Arms: Induction (Main Study + Japan Sub-study): I-SD; Maintenance (Main Study + Japan Sub-study): M-SD; Maintenance (Main Study): TDM Regimen

SUMMARY:
To evaluate safety and efficacy of two adalimumab dosing regimens for induction and maintenance (standard and higher dosing) in achieving clinical remission in subjects with moderately to severely active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative Colitis (UC) for at least 90 days, confirmed by endoscopy during Screening period.
* Active UC with Mayo Score of 6 to 12 points and endoscopy subscore of 2 to 3 despite concurrent or prior treatment with a full and adequate course, in the opinion of the Investigator, with oral corticosteroids or immunosuppressants or both. Mayo Score is confirmed by central reader.

Exclusion Criteria:

* Subject with Crohn's disease (CD) or indeterminate colitis (IC).
* Current diagnosis of fulminant colitis and/or toxic megacolon.
* Subjects with disease limited to the rectum (ulcerative proctitis) during the screening endoscopy.
* Chronic recurring infections or active tuberculosis (TB).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (173):
- United States (42):
  - Digestive Health Specialists of the Southeast /ID# 127844, Dothan, Alabama
  - Ucsd /Id# 122313, La Jolla, California
  - Rocky Mountain Clinical Resear /ID# 122180, Wheat Ridge, Colorado
  - Medical Research Ctr CT /ID# 122179, Hamden, Connecticut
  - Gastro Florida /ID# 170619, Clearwater, Florida
  - Research Associates of South Florida,LLC /ID# 170309, Miami, Florida
  - Gastroenterology Group Naples /ID# 127806, Naples, Florida
  - Shafran Gastroenterology Ctr /ID# 122320, Winter Park, Florida
  - Atlanta Gastro Assoc /ID# 122336, Atlanta, Georgia
  - Gastro Assoc of Central GA /ID# 122318, Macon, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 122183, Chicago, Illinois
  - University of Chicago /ID# 122302, Chicago, Illinois
  - Carle Foundation Hospital /ID# 135955, Urbana, Illinois
  - Louisiana Research Ctr. LLC /ID# 141655, Shreveport, Louisiana
  - University of Maryland Med Ctr /ID# 169734, Baltimore, Maryland
  - MGG Group, Inc.Chevy Chase Clinical Research /ID# 122238, Chevy Chase, Maryland
  - University of Michigan Hospitals /ID# 122240, Ann Arbor, Michigan
  - Mayo Clinic - Rochester /ID# 122244, Rochester, Minnesota
  - Ctr for Digest and Liver Dis /ID# 122182, Mexico, Missouri
  - NYU Langone Long Island CRA /ID# 122177, Great Neck, New York
  - Icahn School of Med Mt. Sinai /ID# 127047, New York, New York
  - Charlotte Gastro Hepatology /ID# 122235, Charlotte, North Carolina
  - Wake Research Associates, LLC /ID# 122157, Raleigh, North Carolina
  - Consultants for Clinical Res /ID# 122304, Cincinnati, Ohio
  - Dayton Gastroenterology, Inc. /ID# 127804, Englewood, Ohio
  - Gastro United of Tulsa /ID# 125436, Tulsa, Oklahoma
  - The Oregon Clinic- Gastro West /ID# 135273, Portland, Oregon
  - University of Pittsburgh MC /ID# 122331, Pittsburgh, Pennsylvania
  - Erlanger Institute for Clinica /ID# 129009, Chattanooga, Tennessee
  - Gastro One /ID# 122339, Germantown, Tennessee
  - Vanderbilt Univ Med Ctr /ID# 125496, Nashville, Tennessee
  - DHAT Research Institute /ID# 170616, Garland, Texas
  - Biopharma Informatic Research /ID# 171150, Houston, Texas
  - Austin Center for Clinical Research /ID# 125396, Pflugerville, Texas
  - Texas Digestive Disease Consul /ID# 141677, Southlake, Texas
  - Texas Digestive Disease Consul /ID# 141678, Southlake, Texas
  - Advanced Research Institute /ID# 126147, Ogden, Utah
  - University of Utah /ID# 122333, Salt Lake City, Utah
  - New River Valley Research Inst /ID# 127801, Christiansburg, Virginia
  - University of Washington /ID# 169721, Seattle, Washington
  - WI Center for Advanced Res /ID# 122178, Milwaukee, Wisconsin
  - Froedtert & the Medical College of Wisconsin /ID# 122261, Milwaukee, Wisconsin
- Austria (5):
  - KH der Elisabethinen Linz GmbH /ID# 127184, Linz, Upper Austria
  - Medizinische Universitat Wien /ID# 127186, Vienna, Vienna
  - Ordination Hainburg an der Don /ID# 127185, Hainburg an der Donau
  - Universitaetsklinik fuer Innere Medizin 1 /ID# 125944, Salzburg
  - KH der Barmherzigen Brueder /ID# 127183, Sankt Veit an der Glan
- Belgium (3):
  - AZ Sint-Lucas /ID# 127187, Ghent
  - UZ Leuven /ID# 126739, Leuven
  - CHU de Liege /ID# 126740, Liège
- Canada (8):
  - University of Calgary /ID# 125715, Calgary, Alberta
  - Zeidler Ledcor Centre /ID# 125713, Edmonton, Alberta
  - Winnipeg Regional Health Autho /ID# 125712, Winnipeg, Manitoba
  - Qe Ii Hsc /Id# 127045, Halifax, Nova Scotia
  - London Health Sciences Centre /ID# 127055, London, Ontario
  - Mount Sinai Hosp.-Toronto /ID# 126590, Toronto, Ontario
  - Toronto Digestive Disease Asso /ID# 127075, Vaughan, Ontario
  - McGill Univ HC /ID# 127046, Montreal, Quebec
- Czechia (2):
  - Hepato-Gastroenterologie HK s.r.o. /ID# 127188, Hradec Králové
  - ISCARE a.s. /ID# 127837, Prague
- Denmark (2):
  - Herlev Hospital /ID# 127191, Herlev, Capital Region
  - Regionhospital Silkeborg /ID# 127190, Silkeborg
- France (10):
  - CHRU Lille - Hôpital Claude Huriez /ID# 127197, Lille, Hauts-de-France
  - CHU NANCY - Hôpital Brabois Adultes /ID# 127196, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU Amiens Picardie /ID# 127194, Amiens, Somme
  - CHU Estaing /ID# 127848, Clermont-Ferrand
  - CHU Dijon /ID# 127861, Dijon
  - CHU de Grenoble - Albet Michal /ID# 127195, Grenoble
  - CHU Saint ELOI /ID# 169007, Montpellier
  - CHU de Nice /ID# 127193, Nice
  - CHU de Saint-Etienne, Hopital Nord /ID# 134490, Saint-Etienne
  - Hopital Rangueil /ID# 127192, Toulouse
- Germany (11):
  - Universitatsklinik Regensburg /ID# 201265, Regensburg, Bavaria
  - Universitatsklinikum Frankfurt /ID# 170300, Frankfurt am Main, Hesse
  - Univ Hosp Schleswig-Holstein, Campus Kiel, Klinik furer Innere Medizin /ID# 127199, Kiel, Schleswig-Holstein
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum /ID# 127203, Berlin
  - Mross, Berlin, DE /ID# 127201, Berlin
  - Gastrostudien GbR /ID# 169246, Berlin
  - Asklepios Westklinikum Hamburg /ID# 127198, Hamburg
  - Universitaetsklinikum Jena /ID# 127205, Jena
  - EUGASTRO GmbH /ID# 127202, Leipzig
  - Universitatsklinikum Magdeburg /ID# 127200, Magdeburg
  - Gastro Campus Research GbR /ID# 126743, Münster
- Hungary (4):
  - Pecsi Tudomanyegyetem Klinikai Kozpont I. sz. Belgyogyaszati Klinika /ID# 127209, Pécs, Pecs
  - Magyar Elhizastudomanyi KKft. /ID# 126589, Budapest
  - Pannonia Maganorvosi Centrum Kft. /ID# 127207, Budapest
  - Szegedi Tudomanyegyetem /ID# 127208, Szeged
- Israel (5):
  - Rabin Medical Center /ID# 127212, Petakh Tikva, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 201365, Tel Aviv, Tel Aviv
  - Soroka University Medical Center /ID# 127213, Beersheba
  - Hadassah University Hospital /ID# 127211, Jerusalem
  - Kaplan Medical Center /ID# 127210, Rehovot
- Italy (10):
  - A.O.U. Policlinico S.Orsola-Malpighi /ID# 129322, Bologna, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini /ID# 127216, Rome, Lazio
  - Policlinico Agostino Gemelli /ID# 127217, Rome, Lazio
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 127138, Milan, Lombardy
  - IBD Center - IRCCS Istituto Clinico Humanitas /ID# 127215, Rozzano, Milano
  - Azienda Ospedaliera Spedali Civili /ID# 127236, Brescia
  - Universita di Padova /ID# 127214, Padua
  - Ospedali Riuniti Villa Sofia-C /ID# 129323, Palermo
  - Policlinico Univ Tor Vergata /ID# 129321, Rome
  - IRCCS Casa Sollievo /ID# 127811, San Giovanni Rotondo
- Japan (24):
  - Yokoyama IBD Clinic /ID# 151560, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 124517, Nagoya, Aichi-ken
  - Toho University Sakura Medical Center /ID# 124497, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital /ID# 124155, Chikushino-shi, Fukuoka
  - Kyushu University Hospital /ID# 124495, Fukuoka, Fukuoka
  - Hidaka Clinic of Coloproctology /ID# 125477, Kurume, Fukuoka
  - Kurume University Hospital /ID# 125275, Kurume-shi, Fukuoka
  - Hiroshima University Hospital /ID# 124496, Hiroshima, Hiroshima
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 124480, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 127836, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 127539, Nishinomiya-shi, Hyōgo
  - Kitasato University Hospital /ID# 137694, Sagamihara-shi, Kanagawa
  - COLO-PROCTOLOGY CENTER Matsushima Clinic /ID# 148423, Yokohama, Kanagawa
  - Susaki Kuroshio Hospital /ID# 125202, Susaki-shi, Kochi
  - Japanese Red Cross Kyoto Daiichi Hos /ID# 127540, Kyoto, Kyoto
  - Osaka Medical College Hospital /ID# 126451, Takatsuki-shi, Osaka
  - Saitama Medical Center /ID# 128875, Kawagoe-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 127675, Ōtsu, Shiga
  - Hamamatsu South Hospital /ID# 124481, Hamamatsu, Shizuoka
  - Medical Hospital of Tokyo Medical and Dental University /ID# 128315, Bunkyo-ku, Tokyo
  - Kitasato Univ Kitasato Inst Ho /ID# 127001, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 148184, Mitaka-shi, Tokyo
  - Wakayama Medical University /ID# 124635, Wakayama, Wakayama
  - Tokyo Yamate Medical Center /ID# 125201, Tokyo
- Academisch Medisch Centrum /ID# 126741, Amsterdam, North Holland, Netherlands
- Poland (12):
  - Szpital Uniwersytecki Nr 2 im. dr J.Biziela w Bydgoszczy /ID# 127141, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Zdrowia MDM /ID# 170303, Warsaw, Masovian Voivodeship
  - Endoterapia PFG Sp. z.o.o. /ID# 126513, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 170301, Gdynia, Pomeranian Voivodeship
  - NZOZ All-Medicus /ID# 128740, Katowice, Silesian Voivodeship
  - H-T.Centrum Medyczne-Endoterapia /ID# 170305, Tychy, Silesian Voivodeship
  - Centrum Medyczne LukaMed Joanna Luka /ID# 170302, Chojnice
  - Centrum Medyczne Sw. Lukaza /ID# 126515, Częstochowa
  - Centrum Diagnostyczno Lecznicze Barska /ID# 170304, Lodz
  - KO-Med Centra Kliniczne Pulawy /ID# 127219, Puławy
  - NZOZ Vivamed /ID# 127218, Warsaw
  - C.M. Szpital Swietej Rodziny /ID# 127838, Lodz, Łódź Voivodeship
- Romania (6):
  - Institutul Clinic Fundeni /ID# 127839, Sector 2, București
  - CMDTA Neomed SRL /ID# 127142, Brasov
  - Spitalul Clinic Judetean de Urgenta /ID# 125418, Cluj-Napoca
  - Tvm Med Serv Srl /Id# 127221, Cluj-Napoca
  - Cabinet Medical Dr. Fratila SRL, Specialitatea Medicina Interna /ID# 127002, Oradea
  - Salvo-San-Ciobanca SRL /ID# 127140, Zalău
- Slovakia (3):
  - Gastroenterologicke centrum ASSIDUO a IBD centrum /ID# 127222, Bratislava
  - Gastroenterologicka Ambulancia /ID# 125632, Bratislava
  - Vseobecna Nemocnica s poliklinikou Lucenec /ID# 127322, Lučenec
- Spain (10):
  - Hospital General Universitario de Alicante /ID# 129261, Alicante
  - Hospital Clinic de Barcelona /ID# 138147, Barcelona
  - Complejo Hospitalario Universitario de Ferrol /ID# 127840, Ferrol
  - Hospital Univ Dr. Negrin /ID# 127841, Las Palmas de Gran Canaria
  - Hospital Univ de la Princesa /ID# 135828, Madrid
  - Hospital General Universitario Gregorio Maranon /ID# 127224, Madrid
  - Hosp Univ 12 de Octubre /ID# 129257, Madrid
  - Hospital Universitario La Paz /ID# 127223, Madrid
  - Hosp Clin Univ de Valencia /ID# 170306, Valencia
  - Hosp Clin Univ Lozano Blesa /ID# 129255, Zaragoza
- Switzerland (2):
  - Kantonsspital St. Gallen /ID# 127843, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich /ID# 127842, Zurich, Canton of Zurich
- Ukraine (5):
  - GI National Institute of Therapy named by L.T. Malaya /ID# 127231, Kharkiv, Kharkivs’ka Oblast’
  - Public Institution Kherson City Clinical Hospital named after le.le. Karabelesh /ID# 127233, Kherson
  - Municipal Clinical Hospital #8 /ID# 127235, Kiev
  - Lviv City Clinical Hospital NO.4 /ID# 127232, Lviv
  - CNPE City Hospital No.6 of Zaporizhzhia City Counsil /ID# 127137, Zaporizhzhia
- United Kingdom (8):
  - Royal Hampshire County Hosp /ID# 169250, Winchester, Hampshire
  - Norfolk and Norwich Univ Hosp /ID# 127139, Norwich, Norfolk
  - Western General Hospital /ID# 204801, Edinburgh
  - St. Mark's Hospital /ID# 127226, Harrow
  - Hull and East Yorkshire Hospitals NHS Trust /ID# 127225, Hull
  - Oxford University Hospitals NHS Foundation Trust The John Radcliffe Hospital /ID# 129324, Oxford
  - Southampton General Hospital /ID# 127228, Southampton
  - The Royal Wolverhampton NHS Tr /ID# 127227, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Reppell M, Zheng X, Dreher I, Blaes J, Regan E, Haslberger T, Guay H, Pivorunas V, Smaoui N. HLA-DQA1*05 Associates With Anti-Tumor Necrosis Factor Immunogenicity and Low Adalimumab Trough Concentrations in Inflammatory Bowel Disease Patients From the SERENE Ulcerative Colitis and Crohn's Disease Studies. J Crohns Colitis. 2025 Jan 11;19(1):jjae129. doi: 10.1093/ecco-jcc/jjae129. PMID 39162746
- [Derived] Verstockt B, Pivorunas V, Al Mahi N, Smaoui N, Guay H, Kennedy NA, Goodhand JR, Lin S, Bai BYH, Hanauer SB, Ferrante M, Panes J, Vermeire S. Baseline TREM-1 Whole Blood Gene Expression Does Not Predict Response to Adalimumab Treatment in Patients with Ulcerative Colitis or Crohn's Disease in the SERENE Studies. J Crohns Colitis. 2024 Apr 23;18(4):493-505. doi: 10.1093/ecco-jcc/jjad170. PMID 37801628
- [Derived] Ponce-Bobadilla AV, Stodtmann S, Chen MJ, Winzenborg I, Mensing S, Blaes J, Haslberger T, Laplanche L, Dreher I, Mostafa NM. Assessing the Impact of Immunogenicity and Improving Prediction of Trough Concentrations: Population Pharmacokinetic Modeling of Adalimumab in Patients with Crohn's Disease and Ulcerative Colitis. Clin Pharmacokinet. 2023 Apr;62(4):623-634. doi: 10.1007/s40262-023-01221-x. Epub 2023 Mar 11. PMID 36905528
- [Derived] Greener T, Boland K, Milgrom R, Ben-Bassat O, Steinhart AH, Silverberg MS, Narula N. Higher adalimumab maintenance regimen is more effective than standard dose in anti-TNF experienced Crohn's disease patients. Eur J Gastroenterol Hepatol. 2021 Oct 1;33(10):1274-1279. doi: 10.1097/MEG.0000000000002250. PMID 34402466
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a Main Study (120 sites in 19 countries) and a Japan Sub-Study (22 sites in Japan).
  After a 3-week screening period, participants were randomized 3:2 to an 8-week double-blind (DB) Induction Period with 2 adalimumab dosing regimens (Induction Standard Dose [I-SD] or Induction Higher Dose [I-HD]).
Pre-assignment Details: At Week 8, participants in Main Study were re-randomized (2:2:1) into 44-week DB Maintenance Period with 3 adalimumab dosing regimens (M-SD, M-HD, or an exploratory Therapeutic Drug Monitoring [TDM] Regimen). Participants in Japan Sub-study were re-randomized (1:1) into 44-week DB Maintenance Period with 2 adalimumab dosing regimens (M-SD, M-HD).
Groups:
- Induction (Main Study + Japan Sub-study): I-SD: Induction Standard Dose (I-SD): Double-blind adalimumab regimen of 160 mg at Week 0 followed by 80 mg at Week 2, 40 mg at Week 4, and 40 mg at Week 6.
- Induction (Main Study + Japan Sub-study): I-HD: Induction Higher Dose (I-HD): Double-blind adalimumab regimen of 160 mg at Weeks 0, 1, 2, and 3 followed by 40 mg at Week 4 and 40 mg at Week 6.
- Maintenance (Main Study + Japan Sub-study): M-SD: Maintenance Standard Dose (M-SD): Double-blind adalimumab 40 mg every other week (eow), for 44 weeks.
- Maintenance (Main Study + Japan Sub-study): M-HD: Maintenance Higher Dose (M-HD): Double-blind adalimumab 40 mg every week (ew) for 44 weeks.
- Maintenance (Main Study): TDM Regimen: Exploratory Therapeutic Drug Monitoring (TDM) Regimen: Double-blind adalimumab 40 mg eow at Week 8 and Week 10, with possible dose adjustments at Weeks 12, 24, and 37 based on criteria assessing blinded adalimumab serum concentration and rectal bleeding subscore assessments.
Period: Induction Study
Arm/Group | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD | Maintenance (Main Study): TDM Regimen
Started | 379 | 573 | 0 | 0 | 0
Enrolled in Main Study | 340 | 512 | 0 | 0 | 0
Enrolled in Japan Sub-Study | 39 | 61 | 0 | 0 | 0
Completed | 332 | 514 | 0 | 0 | 0
Not Completed | 47 | 59 | 0 | 0 | 0
Not completed — Adverse Event | 13 | 19 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 22 | 27 | 0 | 0 | 0
Not completed — Requires Alternative/Prohibited Therapy | 4 | 5 | 0 | 0 | 0
Not completed — Subject Noncompliance | 1 | 1 | 0 | 0 | 0
Not completed — Other, Not Specified | 3 | 2 | 0 | 0 | 0
Period: Maintenance Study
Arm/Group | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD | Maintenance (Main Study): TDM Regimen
Started | 0 | 0 | 345 | 350 | 151
Completed | 0 | 0 | 221 | 246 | 105
Not Completed | 0 | 0 | 124 | 104 | 46
Not completed — Adverse Event | 0 | 0 | 25 | 22 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 11 | 5 | 7
Not completed — Lost to Follow-up | 0 | 0 | 4 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 70 | 55 | 19
Not completed — Requires Alternative/Prohibited Therapy | 0 | 0 | 7 | 3 | 4
Not completed — Subject Non-Compliance | 0 | 0 | 1 | 3 | 2
Not completed — Other, Not Specified | 0 | 0 | 6 | 14 | 2
Not completed — Unknown Reason | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Induction (Main Study + Japan Sub-study): I-HD: Induction Higher Dose: Double-blind adalimumab regimen of 160 mg at Weeks 0, 1, 2, and 3 followed by 40 mg at Week 4 and 40 mg at Week 6.
- Total: Total of all reporting groups
Arm/Group | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD | Total
Number analyzed (Participants) | 379 | 573 | 952
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (13.14) | 40.5 (12.89) | 40.4 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 239 | 405
  Male | 213 | 334 | 547
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 326 | 484 | 810
  Black or African American | 8 | 16 | 24
  Asian | 44 | 70 | 114
  Native Hawaiian/Other Pacific Islander | 0 | 1 | 1
  Multiracial | 1 | 1 | 2
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 28 | 47
  Japanese | 39 | 61 | 100
  Other, Not Specified | 321 | 484 | 805
Region [Count of Participants; unit: Participants]
  United States | 65 | 113 | 178
  Non-United States | 314 | 460 | 774
Full Mayo Score (FMS) [Mean (Standard Deviation); unit: units on a scale] — The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Population: participants with an assessment
  units on a scale
    number analyzed (Participants) | 379 | 570 | 949
    (all) | 8.69 (1.509) | 8.87 (1.571) | 8.80 (1.548)
FMS: Rectal Bleeding Subscore [Mean (Standard Deviation); unit: units on a scale] — The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Population: participants with an assessment
  units on a scale
    number analyzed (Participants) | 379 | 570 | 949
    (all) | 1.68 (0.955) | 1.75 (0.967) | 1.72 (0.962)

OUTCOME MEASURES:

1. Primary Outcome: Induction Period Primary Endpoint: Percentage of Participants With Clinical Remission Per Full Mayo Score (FMS) at Week 8
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Clinical remission per FMS is defined as Mayo Score ≤ 2 and no individual subscore > 1.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Induction (Main Study): I-SD; Induction (Main Study + Japan Sub-study): I-SD: Induction Standard Dose: Double-blind adalimumab regimen of 160 mg at Week 0 followed by 80 mg at Week 2, 40 mg at Week 4, and 40 mg at Week 6.
- Induction (Main Study): I-HD; Induction (Main Study + Japan Sub-study): I-HD: Induction Higher Dose: Double-blind adalimumab regimen of 160 mg at Weeks 0, 1, 2, and 3 followed by 40 mg at Week 4 and 40 mg at Week 6.
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 10.9 | 13.3 | 11.6 | 13.8
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; Adjusted risk difference, 95% confidence interval for the difference in the proportions between the treatment groups and P-value were calculated using Cochran-Mantel-Haenszel test adjusted for previous infliximab use and baseline corticosteroid use; Test type: Superiority; p = 0.269, Cochran-Mantel-Haenszel; Adjusted risk difference = 2.5, 95% CI 2-sided [-2.0 to 7.0] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; Test type: Superiority; p = 0.447, Breslow-Day test; Breslow-Day test of homogeneity across strata
Statistical Analysis 3: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.301, Cochran-Mantel-Haenszel; Adjusted risk difference = 2.3, 95% CI 2-sided [-2.0 to 6.6] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 4: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; Test type: Superiority; p = 0.502, Breslow-Day test; Breslow-Day test of homogeneity across strata

2. Primary Outcome: Maintenance Period Primary Endpoint: Percentage of Week 8 Responders (Per FMS) With Clinical Remission (Per FMS) at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders (per FMS) are defined as participants with a decrease in Full Mayo score of ≥ 3 points and ≥ 30% from Baseline plus a decrease from baseline in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1. Clinical remission per FMS is defined as Mayo Score ≤ 2 and no individual subscore > 1.
Time Frame: Week 52
Population: ITT-Responder population (I-ITT-RP): all participants in the Induction ITT population who achieve Week 8 response based on the FMS utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, the TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Groups:
- Maintenance (Main Study): M-SD; Maintenance (Main Study + Japan Sub-study): M-SD: Maintenance Standard Dose: Double-blind adalimumab 40 mg every other week (eow), for 44 weeks.
- Maintenance (Main Study): M-HD; Maintenance (Main Study + Japan Sub-study): M-HD: Maintenance Higher Dose: Double-blind adalimumab 40 mg every week (ew) for 44 weeks.
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 145 | 152 | 163 | 175
percentage of participants | 29.0 | 39.5 | 30.1 | 41.1
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; Adjusted risk difference, 95% confidence interval for the difference in the proportions between the treatment groups and P-value were calculated using Cochran-Mantel-Haenszel (CMH) test adjusted for induction treatment regimen and week 8 remission status; Test type: Superiority; p = 0.069, Cochran-Mantel-Haenszel; Adjusted risk difference = 9.9, 95% CI 2-sided [-0.8 to 20.6] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; Test type: Superiority; p = 0.085, Breslow-Day test; Breslow-Day test of homogeneity across strata
Statistical Analysis 3: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.045, Cochran-Mantel-Haenszel; Adjusted risk difference = 10.3, 95% CI 2-sided [0.2 to 20.4] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 4: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; Test type: Superiority; p = 0.106, Breslow-Day test; Breslow-Day test of homogeneity across strata

3. Secondary Outcome: Induction Period Ranked Secondary Endpoint 1: Percentage of Participants With Endoscopic Improvement at Week 8
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 27.1 | 31.1 | 26.9 | 30.5
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.181, Cochran-Mantel-Haenszel; Adjusted risk difference = 4.2, 95% CI 2-sided [-2.0 to 10.5] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.200, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.8, 95% CI 2-sided [-2.0 to 9.7] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

4. Secondary Outcome: Induction Period Ranked Secondary Endpoint 2: Percentage of Participants With Fecal Calprotectin < 150 mg/kg at Week 8
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 27.1 | 31.1 | 26.9 | 30.5
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.300, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.0, 95% CI 2-sided [-2.6 to 8.6] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.254, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.1, 95% CI 2-sided [-2.2 to 8.4] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

5. Secondary Outcome: Induction Period Ranked Secondary Endpoint 3: Percentage of Participants With Inflammatory Bowel Disease Questionnaire (IBDQ) Response (Increase of IBDQ ≥ 16 From Baseline) at Week 8
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). Total IBDQ score is the sum of the responses to the individual IBDQ questions, and ranges from 32 to 224 with higher scores indicating a better quality of life.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 60.9 | 67.2 | 60.7 | 65.3
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.050, Cochran-Mantel-Haenszel; Adjusted risk difference = 6.5, 95% CI 2-sided [-0.0 to 13.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.131, Cochran-Mantel-Haenszel; Adjusted risk difference = 4.8, 95% CI 2-sided [-1.4 to 11.0] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

6. Secondary Outcome: Induction Period Ranked Secondary Endpoint 4: Percentage of Participants With Clinical Response Per FMS at Week 8
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Clinical response is defined as a decrease in FMS of ≥ 3 points and ≥ 30% from baseline, plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 40.0 | 47.1 | 38.8 | 47.3
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.035, Cochran-Mantel-Haenszel; Adjusted risk difference = 7.3, 95% CI 2-sided [0.5 to 14.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Adjusted risk difference = 8.7, 95% CI 2-sided [2.3 to 15.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

7. Secondary Outcome: Induction Period Ranked Secondary Endpoint 5: Percentage of Participants With Endoscopic Remission at Week 8
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Endoscopic remission is defined as an endoscopy subscore of 0.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 10.0 | 13.1 | 10.0 | 12.9
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.160, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.2, 95% CI 2-sided [-1.3 to 7.6] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.166, Cochran-Mantel-Haenszel; Adjusted risk difference = 2.9, 95% CI 2-sided [-1.2 to 7.1] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

8. Secondary Outcome: Induction Period Ranked Secondary Endpoint 6: Percentage of Participants Achieving Response in IBDQ Bowel Symptom Domain at Week 8
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). The range for Bowel Symptom domain score is 10 (severe problem) to 70 (normal health). Response in IBDQ Bowel Symptom domain is defined as an increase of IBDQ Bowel Symptom domain score ≥ 6.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 63.2 | 71.3 | 63.1 | 69.8
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Adjusted risk difference = 8.3, 95% CI 2-sided [1.9 to 14.7] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel; Adjusted risk difference = 7.0, 95% CI 2-sided [0.9 to 13.0] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

9. Secondary Outcome: Induction Period Ranked Secondary Endpoint 7: Percentage of Participants Achieving Response in IBDQ Fatigue Item at Week 8
Description: The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). The IBDQ Fatigue item score range is from 1 (severe problem) to 7 (normal health). Response is defined as an increase of IBDQ Fatigue item score ≥ 1.
Time Frame: Week 8
Population: Induction Study Intent-to-Treat (ITT) set: all participants who were randomized at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Induction (Main Study): I-SD | Induction (Main Study): I-HD | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD
Number analyzed (Participants) | 340 | 512 | 379 | 573
percentage of participants | 57.1 | 61.1 | 57.5 | 59.9
Statistical Analysis 1: Comparison: Induction (Main Study): I-SD vs Induction (Main Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.218, Cochran-Mantel-Haenszel; Adjusted risk difference = 4.2, 95% CI 2-sided [-2.5 to 10.9] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)
Statistical Analysis 2: Comparison: Induction (Main Study + Japan Sub-study): I-SD vs Induction (Main Study + Japan Sub-study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.456, Cochran-Mantel-Haenszel; Adjusted risk difference = 2.4, 95% CI 2-sided [-4.0 to 8.8] — Risk difference = (adalimumab higher induction dose - adalimumab standard induction dose)

10. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 1: Percentage of Week 8 Responders (Per FMS) With Endoscopic Improvement at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders are defined as participants with a decrease in FMS of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 145 | 152 | 163 | 175
percentage of participants | 41.4 | 51.3 | 41.7 | 52.0
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.098, Cochran-Mantel-Haenszel; Adjusted risk difference = 9.5, 95% CI 2-sided [-1.7 to 20.8] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.066, Cochran-Mantel-Haenszel; Adjusted risk difference = 9.9, 95% CI 2-sided [-0.7 to 20.5] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

11. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 2: Percentage of Week 8 Responders With Steroid Usage at Baseline and Steroid Free at Least 90 Days at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders, per FMS, are defined as participants with a decrease in FMS of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 52
Population: I-ITT-RP: participants in the Induction ITT population who achieve Week 8 response based on the FMS utilizing the endoscopy subscore provided by the central reader. Participants with steroid use at Baseline. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 92 | 95 | 103 | 108
percentage of participants | 53.3 | 74.7 | 54.4 | 74.1
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW; Adjusted risk difference = 21.5, 95% CI 2-sided [7.6 to 35.4]
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Adjusted risk difference = 19.7, 95% CI 2-sided [6.6 to 32.7] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

12. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 3: Percentage of Week 8 Responders With Steroid Usage at Baseline and Steroid Free at Least 90 Days and With Clinical Remission at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders, per FMS, are defined as participants with a decrease in FMS of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1. Clinical remission is defined as FMS ≤ 2 with no subscore > 1.
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 92 | 95 | 103 | 108
percentage of participants | 27.2 | 38.9 | 28.2 | 39.8
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.093, Cochran-Mantel-Haenszel; Adjusted risk difference = 11.5, 95% CI 2-sided [-1.9 to 25.0] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.088, Cochran-Mantel-Haenszel; Adjusted risk difference = 11.1, 95% CI 2-sided [-1.7 to 23.8] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

13. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 4: Percentage of Week 8 Remitters (Per FMS) With Clinical Remission (Per FMS) at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 remitters are defined as participants with clinical remission (per FMS) at Week 8. Clinical remission is defined as a FMS ≤ 2 with no subscore > 1. Endoscopy subscore provided by the central reader.
Time Frame: Week 52
Population: ITT-Remitter (ITT-RM) Population included all participants in the ITT population who achieved Week 8 remission based on the FMS utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 37 | 42 | 45 | 52
percentage of participants | 40.5 | 57.1 | 44.4 | 55.8
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.161, Cochran-Mantel-Haenszel; Adjusted risk difference = 15.9, 95% CI 2-sided [-6.3 to 38.2] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.312, Cochran-Mantel-Haenszel; Adjusted risk difference = 10.4, 95% CI 2-sided [-9.8 to 30.6] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

14. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 5: Percentage of Week 8 Remitters (Per FMS) With Endoscopic Improvement at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 remitters are defined as participants with clinical remission (per FMS) at Week 8. Clinical remission is defined as a FMS ≤ 2 with no subscore > 1. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1. Endoscopy subscore provided by the central reader.
Time Frame: Week 52
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 37 | 42 | 45 | 52
percentage of participants | 51.4 | 64.3 | 55.6 | 61.5
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.272, Cochran-Mantel-Haenszel; Adjusted risk difference = 12.3, 95% CI 2-sided [-9.7 to 34.4] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.600, Cochran-Mantel-Haenszel; Adjusted risk difference = 5.3, 95% CI 2-sided [-14.6 to 25.2] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

15. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 6: Percentage of Week 8 Remitters (Per FMS) With Steroid Usage at Baseline and Steroid Free at Least 90 Days at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 remitters are defined as participants with clinical remission (per FMS) at Week 8. Clinical remission is defined as a FMS ≤ 2 with no subscore > 1.
Time Frame: Week 52
Population: ITT-RM Population: participants in ITT population who achieved Week 8 remission based on the FMS utilizing the endoscopy subscore provided by the central reader. Participants with steroid use at Baseline. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 26 | 27 | 32 | 35
percentage of participants | 53.8 | 77.8 | 56.3 | 71.4
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.074, Cochran-Mantel-Haenszel; Adjusted risk difference = 23.8, 95% CI 2-sided [-2.3 to 49.9] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.210, Cochran-Mantel-Haenszel; Adjusted risk difference = 15.0, 95% CI 2-sided [-8.5 to 38.4] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

16. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 7: Percentage of Week 8 Remitters (Per FMS) With Steroid Usage at Baseline and Steroid Free at Least 90 Days and With Clinical Remission (Per FMS) at Week 52
Description: as for outcome 15
Time Frame: Week 52
Population: ITT-RM Population: all participants in the ITT population who achieved Week 8 remission based on the FMS utilizing the endoscopy subscore provided by the central reader. Participants with steroid usage. Non-responder imputation. Per protocol, the TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 26 | 27 | 32 | 35
percentage of participants | 34.6 | 55.6 | 37.5 | 51.4
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.151, Cochran-Mantel-Haenszel; Adjusted risk difference = 20.0, 95% CI 2-sided [-7.3 to 47.3] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.299, Cochran-Mantel-Haenszel; Adjusted risk difference = 12.8, 95% CI 2-sided [-11.3 to 36.8] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

17. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 8: Percentage of Week 8 Responders (Per FMS) With IBDQ Response (Increase of IBDQ ≥ 16 From Baseline) at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders are defined as participants with a decrease in FMS of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1. The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). Total IBDQ score is the sum of responses to the individual IBDQ questions, and ranges from 32 to 224 with higher scores indicating a better quality of life.
Time Frame: Week 52
Population: ITT-Responder population (ITT-RP): all participants in the Induction ITT population who achieve Week 8 response based on the FMS utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, the TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 145 | 152 | 163 | 175
percentage of participants | 62.1 | 66.4 | 62.6 | 65.7
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.422, Cochran-Mantel-Haenszel; Adjusted risk difference = 4.5, 95% CI 2-sided [-6.4 to 15.3] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.513, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.4, 95% CI 2-sided [-6.8 to 13.6] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

18. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 9: Percentage of Week 8 Non-Responders With Clinical Remission (Per FMS) at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 non-responders are defined as participants not meeting the criteria of response (defined as a decrease in FMS of ≥ 3 points and ≥ 30% from baseline, plus a decrease in the rectal bleeding subscore [RBS] ≥ 1 or an absolute RBS ≤ 1) at Week 8. Clinical remission is defined as a FMS ≤ 2 with no subscore > 1.
Time Frame: Week 52
Population: ITT-Non-Responder (ITT-NRP) Population: all participants in ITT who did not achieve Week 8 response based on the Full Mayo Score utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 157 | 152 | 182 | 175
percentage of participants | 12.1 | 15.8 | 12.1 | 16.0
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.351, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.7, 95% CI 2-sided [-4.1 to 11.4] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.292, Cochran-Mantel-Haenszel; Adjusted risk difference = 3.9, 95% CI 2-sided [-3.3 to 11.1] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

19. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 10: Percentage of Week 8 Non-Remitters With Clinical Remission (Per FMS) at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 non-remitters are defined as participants not meeting the criteria of clinical remission at Week 8. Clinical remission is defined as a FMS ≤ 2 with no subscore > 1.
Time Frame: Week 52
Population: ITT-Non-Remitter (ITT-NRM) Population: all participants in ITT who did not achieve Week 8 remission based on the FMS utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 265 | 262 | 300 | 298
percentage of participants | 17.4 | 22.9 | 17.0 | 23.8
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.121, Cochran-Mantel-Haenszel; Adjusted risk difference = 5.4, 95% CI 2-sided [-1.4 to 12.1] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.046, Cochran-Mantel-Haenszel; Adjusted risk difference = 6.5, 95% CI 2-sided [0.1 to 12.8] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

20. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 11: Percentage of Week 8 Responders (Per FMS) With Endoscopic Subscore of 0 at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders (per Full Mayo score) are defined as participants with a decrease in Full Mayo score of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1. Endoscopic remission is defined as an endoscopy subscore of 0.
Time Frame: Week 52
Population: ITT-RP: participants in the Induction ITT population who achieve Week 8 response based on the FMS utilizing the endoscopy subscore provided by the central reader. Participants who were remitters at Week 8. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 145 | 152 | 163 | 175
percentage of participants | 27.6 | 35.5 | 27.0 | 35.4
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.159, Cochran-Mantel-Haenszel; Adjusted risk difference = 7.5, 95% CI 2-sided [-2.9 to 17.9] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.109, Cochran-Mantel-Haenszel; Adjusted risk difference = 8.0, 95% CI 2-sided [-1.8 to 17.9] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

21. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 12: Percentage of Week 8 Remitters (Per FMS) With Endoscopic Subscore of 0 at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 remitters are defined as participants with clinical remission (per FMS) at Week 8. Clinical remission is defined as a FMS ≤ 2 with no subscore > 1. Endoscopic remission is defined as an endoscopy subscore of 0.
Time Frame: Week 52
Population: ITT-Remitter (ITT-RM) Population: all participants in ITT who achieved Week 8 remission based on the Full Mayo Score utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 37 | 42 | 45 | 52
percentage of participants | 45.9 | 47.6 | 42.2 | 44.2
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.903, Cochran-Mantel-Haenszel; Adjusted risk difference = 1.4, 95% CI 2-sided [-21.0 to 23.8] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.901, Cochran-Mantel-Haenszel; Adjusted risk difference = 1.3, 95% CI 2-sided [-18.8 to 21.3] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

22. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 13: Percentage of Week 8 Responders (Per FMS) With Response in IBDQ Bowel Symptom Domain at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders are defined as participants with a decrease in FMS of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore [RBS] ≥ 1 or an absolute RBS ≤ 1. The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). Bowel Symptom domain score range is 10 (severe problem) to 70 (normal health). Response is defined as increase of Bowel Symptom domain score ≥ 6 from baseline.
Time Frame: Week 52
Population: ITT-Responder population (ITT-RP): all participants in the Induction ITT population who achieve Week 8 response based on the FMS utilizing the endoscopy subscore provided by the central reader. Non-responder imputation. Per protocol, TDM Regimen arm was used to analyze exploratory outcome measures only (and therefore is not included).
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 145 | 152 | 163 | 175
percentage of participants | 62.1 | 69.7 | 62.6 | 71.4
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.160, Cochran-Mantel-Haenszel; Adjusted risk difference = 7.7, 95% CI 2-sided [-3.0 to 18.4] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.076, Cochran-Mantel-Haenszel; Adjusted risk difference = 9.1, 95% CI 2-sided [-0.9 to 19.1] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

23. Secondary Outcome: Maintenance Period Ranked Secondary Endpoint 14: Percentage of Week 8 Responders (Per FMS) With Response in IBDQ Fatigue Item at Week 52
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Negative changes indicate improvement. Week 8 responders are defined as participants with a decrease in FMS of ≥ 3 points and ≥ 30% from Baseline plus a decrease in the rectal bleeding subscore (RBS) ≥ 1 or an absolute RBS ≤ 1. The IBDQ is a self-administered 32-item questionnaire to evaluate quality of life across 4 dimensional scores: bowel, systemic, social and emotional. Responses to each question range from 1 (severe problem) to 7 (normal health). Response in IBDQ fatigue item (range 1 [severe problem] to 7 [normal health]) is defined as increase of IBDQ fatigue item ≥ 1 from baseline.
Time Frame: Week 52
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance (Main Study): M-SD | Maintenance (Main Study): M-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD
Number analyzed (Participants) | 145 | 152 | 163 | 175
percentage of participants | 53.8 | 61.2 | 55.2 | 59.4
Statistical Analysis 1: Comparison: Maintenance (Main Study): M-SD vs Maintenance (Main Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.207, Cochran-Mantel-Haenszel; Adjusted risk difference = 7.3, 95% CI 2-sided [-4.0 to 18.6] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW
Statistical Analysis 2: Comparison: Maintenance (Main Study + Japan Sub-study): M-SD vs Maintenance (Main Study + Japan Sub-study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.440, Cochran-Mantel-Haenszel; Adjusted risk difference = 4.2, 95% CI 2-sided [-6.4 to 14.8] — Risk difference = Adalimumab 40mg EW - Adalimumab 40mg EOW

ADVERSE EVENTS:
Time Frame: See time frame specifics detailed for each reporting group in their respective descriptions below. Participants were contacted 70 days following study drug discontinuation for an assessment of any new or ongoing adverse events, except those participants who continued on adalimumab therapy after the end of study participation.
Description: Treatment-emergent adverse events (TEAEs) are presented.
Groups:
- Induction (Main Study + Japan Sub-study): I-SD: Induction Standard Dose: Double-blind adalimumab regimen of 160 mg at Week 0 followed by 80 mg at Week 2, 40 mg at Week 4, and 40 mg at Week 6.
  TEAEs during induction period: events with an onset date on or after first dose date of study drug in induction period and up to 70 days after last dose date of the study drug in induction period and prior to first dose date of study drug in maintenance period. Mean duration of treatment was 57.5 days.
- Induction (Main Study + Japan Sub-study): I-HD: Induction Higher Dose: Double-blind adalimumab regimen of 160 mg at Weeks 0, 1, 2, and 3 followed by 40 mg at Week 4 and 40 mg at Week 6.
  TEAEs during induction period: events with an onset date on or after first dose date of study drug in induction period and up to 70 days after last dose date of the study drug in induction period and prior to first dose date of study drug in maintenance period. Mean duration of treatment was 55.0 days.
- Maintenance (Main Study + Japan Sub-study): M-SD: Maintenance Standard Dose: Double-blind adalimumab 40 mg every other week (eow), for 44 weeks.
  TEAEs during maintenance period: events with an onset date on or after first dose date of study drug in maintenance period and up to 70 days after the last dose date of the study drug in maintenance period. Mean duration of treatment was 251.5 days.
- Maintenance (Main Study + Japan Sub-study): M-HD: Maintenance Higher Dose: Double-blind adalimumab 40 mg every week (ew) for 44 weeks.
  TEAEs during maintenance period: events with an onset date on or after first dose date of study drug in maintenance period and up to 70 days after the last dose date of the study drug in maintenance period. Mean duration of treatment was 263.1 days.
- Maintenance (Main Study): TDM Regimen: Double-blind adalimumab 40 mg eow at Week 8 and Week 10, with possible dose adjustments at Weeks 12, 24, and 37 based on criteria assessing blinded adalimumab serum concentration and rectal bleeding subscore (RBS) assessments.
  TEAEs during maintenance period: events with an onset date on or after first dose date of study drug in maintenance period and up to 70 days after the last dose date of the study drug in maintenance period. Mean duration of treatment was 255.9 days.
Arm/Group | Induction (Main Study + Japan Sub-study): I-SD | Induction (Main Study + Japan Sub-study): I-HD | Maintenance (Main Study + Japan Sub-study): M-SD | Maintenance (Main Study + Japan Sub-study): M-HD | Maintenance (Main Study): TDM Regimen
All-Cause Mortality (participants affected / at risk) | 2/379 | 4/573 | 2/345 | 2/350 | 0/151
Serious Adverse Events (participants affected / at risk) | 19/379 | 22/573 | 44/345 | 44/350 | 15/151
Other Adverse Events (participants affected / at risk) | 74/379 | 112/573 | 140/345 | 141/350 | 47/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (Main Study + Japan Sub-study): I-SD (N=379) | Induction (Main Study + Japan Sub-study): I-HD (N=573) | Maintenance (Main Study + Japan Sub-study): M-SD (N=345) | Maintenance (Main Study + Japan Sub-study): M-HD (N=350) | Maintenance (Main Study): TDM Regimen (N=151)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (2) | 3 (4) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OPTIC ATROPHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANOGENITAL DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 12 (17) | 13 (13) | 16 (16) | 18 (21) | 6 (6)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PORTOSPLENOMESENTERIC VENOUS THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXTERNAL EAR CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERINEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STERNITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TUBERCULOSIS OF INTRATHORACIC LYMPH NODES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VARICELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FIBROMATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC INFLAMMATORY DEMYELINATING POLYRADICULONEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MONONEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BINGE DRINKING (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
SINUS POLYP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EXCESSIVE SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LINEAR IGA DISEASE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBCORNEAL PUSTULAR DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WOUND DRAINAGE (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (Main Study + Japan Sub-study): I-SD (N=379) | Induction (Main Study + Japan Sub-study): I-HD (N=573) | Maintenance (Main Study + Japan Sub-study): M-SD (N=345) | Maintenance (Main Study + Japan Sub-study): M-HD (N=350) | Maintenance (Main Study): TDM Regimen (N=151)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 20 (22) | 18 (18) | 60 (70) | 47 (58) | 23 (29)
NASOPHARYNGITIS (Infections and infestations) | 16 (18) | 29 (34) | 47 (61) | 46 (57) | 11 (20)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 6 (6) | 22 (25) | 19 (20) | 9 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (11) | 18 (19) | 23 (27) | 23 (27) | 5 (5)
HEADACHE (Nervous system disorders) | 23 (32) | 48 (62) | 17 (19) | 22 (36) | 8 (9)
RASH (Skin and subcutaneous tissue disorders) | 11 (11) | 10 (10) | 11 (13) | 20 (24) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02065622/SAP_001.pdf
  • Study Protocol (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT02065622/Prot_002.pdf